CLINICAL TRIAL: NCT04938206
Title: DIStinguishing ChildrEn at Low Risk of Severe infectioN in Case of Febrile Neutropenia-7: Impact Study of a Clinical Decision Rule
Acronym: DISCERN-FN7
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the difficulties encountered in including
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018_99; 2019-A01025-52 (Other: ID-RCB number,ANSM); PREPS-18-0507 (Other: DGOS number)
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Neutropenia, Febrile
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- management reduction strategy (Experimental): Patients classified as low risk by the DRC who will have a reduction in the management of their post-chemotherapy NF.
  Interventions: Procedure: The Clinical Decision Rule
- standard management (Active Comparator): Patients classified as low risk by the DRC who will have standard management of post-chemotherapy NF.
  Interventions: Procedure: The Clinical Decision Rule

INTERVENTIONS:
Procedure: The Clinical Decision Rule — The Clinical Decision Rule will be applied to all patients included in the study at different times depending on the type of cancer: at H12-H24 of admission for patients with solid tumor; at H24-H48 for patients with hematological cancer. Patients classified as being at low risk of severe infection by the DRC were then randomized to a control group under standard management or to an experimental group with therapeutic relief. Treatment reduction for the experimental group was started immediately after randomization, in hospital. Discharge was proposed 24 hours later, with follow-up every two days, by telephone or in

SUMMARY:
Febrile neutropenia (NF) is the leading cause of unscheduled hospitalization in children with cancer. Management classically involves emergency admission to hospital for intravenous antibiotic treatment until resolution of fever and neutropenia. However, children with NF are a heterogeneous group with varying risks of severe infection (10-29%). This approach, which is recognized as excessive for low-risk episodes of severe infection, particularly in terms of quality of life and cost, is no longer recommended. Management should move to a more personalized model that takes into account the individual probability of severe infection. Clinical decision rules (CDRs) have been proposed to facilitate risk stratification, but none are useful in our French population because of insufficient reproducibility or effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Followed for hemopathy or cancer,
* Presenting with post-chemotherapy NF,
* With social security coverage,
* With parents able to provide appropriate home supervision,
* Consent of parents and child if able to give consent.

Exclusion Criteria:

* NF to diagnosis of tumor disease,
* Child with palliative care,
* Child who has had an allogeneic hematopoietic stem cell transplant within the past year,
* NF immediately following an autologous hematopoietic stem cell transplant,
* Participation in the study during a previous NF,
* Curative antibiotic therapy or documented infection prior to admission,
* Initial management at a non-investigative center,
* Refusal of the child or parents to participate

Translated with www.DeepL.com/Translator (free version)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Change in quality of life score, calculated from the PedsQL™ scale between inclusion and Day 6. | at day 6
  The Pediatric Quality of Life Inventory (PedsQL) is a brief measure of health-related quality of life in children and young people. The measure can be completed by parents (the Proxy Report) as well as children and young people (the Self-Report).
  On the PedsQL Generic Core Scales, for ease of interpretability, items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life).
  To reverse score, transform the 0-4 scale items to 0-100 as follows: 0=100, 1=75, 2=50, 3=25, 4=0.

CONTACTS AND LOCATIONS:
Overall Officials: François Dubos, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France